CLINICAL TRIAL: NCT01410929
Title: Evaluation of Vertebral Compression Fracture Fixation With RF Kyphoplasty in Patients With Multiple Myeloma
Acronym: MM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: DFINE Inc. (Industry)
Responsible Party: Frank D. Vrionis MD, MPH, PhD, H. Lee Moffitt Cancer Center
Organization: Merit Medical Systems, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-10-001
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Myeloma; Compression Fracture of Vertebral Column
Keywords: multiple myeloma; VCF; Vertebral Compression Fracture; Spine; Kyphoplasty; Back pain; Cancer
MeSH Terms: conditions — Multiple Myeloma; Back Pain; Neoplasms | interventions — Kyphoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Kyphoplasty/Vertebral Augmentation (Device-StabiliT) — Targeted Vertebral Augmentation for the treatment of pathological fractures of the spine caused by multiple myeloma
  Other Names: Targeted Vertebral Augmentation; Kyphoplasty

SUMMARY:
The objective of this post market clinical study is to collect prospective clinical data to confirm the efficacy of RF Kyphoplasty for the treatment of pathological fractures of the spine caused by multiple myeloma.

DETAILED DESCRIPTION:
Myeloma is the commonest primary cancer affecting the spine. Painful vertebral compression fractures (VCFs) affect approximately 30% of myeloma patients. As myeloma patients live longer, it is especially relevant to provide the best available treatment for pain and reduce disabilities that can result from VCFs.

Cement delivery is a well established treatment method for treating painful vertebrae compromised by tumor and/or osteoporosis. The StabiliT Vertebral Augmentation System (DFine Inc.) is a unique percutaneous vertebral augmentation system designed to provide the physician a means of creating targeted cavities and an ultra-high viscosity cement (using RF Energy) that can be delivered over an extended period of time in order to allow for controlled, targeted vertebral augmentation in multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of multiple myeloma and evidence of myelomatous lesions in the spine, including plasmacytomas, lytic lesions and fractures.
2. One to 6 painful (pain on palpation/percussion over fractured vertebral body) VCF(s), T3-L5, with bone marrow edema imaged by magnetic resonance imaging (MRI) (Subjects with 4-6 fractures treatment will be divided into two sessions 1- 7 days apart)
3. History of fracture related pain less than ≤ 3 months old
4. Pain VAS score ≥4 on a scale of 0 to 10. When the subject is newly diagnosed with multiple myeloma, the pain assessment must not be done until after completion of at least one pulse of steroid therapy or one week after the initiation of active multiple myeloma chemotherapy. Pain represents worst pain without use of narcotic medications.
5. Roland Morris Disability Questionnaire score ≥ 10 on 0 to 24 scale
6. Subjects is ≥ 21 years old.
7. No change in chemotherapy regimen (change in dose(s) permitted) for 1 month prior to enrollment
8. No change in chemotherapy regimen (change in dose(s) permitted) planned for at least 1 month following enrollment
9. Subject has no major surgery to the spine planned for at least 1 month following enrollment
10. Subject has sufficient mental capacity to comply with the protocol requirements
11. Subject must be willing and able to comply with specified follow-up evaluations
12. Subject understands the potential risks and benefits of participating in the study and is willing to provide written informed consent.
13. Female subjects must either be no longer capable of reproduction or taking acceptable measures to prevent pregnancy during the study

Exclusion Criteria:

1. Subjects with primary tumors of the bone (e.g., osteosarcoma) or osteoblastic metastases at site of the index VCF. Subjects with these tumors in anatomic sites other than the index VCF are eligible.
2. Subject is concurrent Phase I investigational anti-cancer treatment
3. Subject has significant clinical morbidities (aside from the index fracture(s) and cancer) that may potentially interfere with the collection of data concerning pain and function
4. Subject has VCF morphology deemed unsuitable for RF Kyphoplasty (e.g. vertebral planna)
5. Additional non-kyphoplasty surgical treatment is required for the index fracture
6. Subjects requiring the use of high-dose steroid (≥ 100 mg prednisone or 20 mg dexamethasone per day), intravenous (IV) pain medication, or nerve block to control chronic back pain unrelated to index VCF(s). Subjects who receive high-dose steroids for treatment of their cancer (for at least 30 days) are eligible.
7. Subjects with a platelet count of < 20,000
8. Subject has spinal cord compression or significant canal compromise requiring decompression
9. Subjects with VCFs due to osteoporosis
10. Subject has medical/surgical conditions contrary to the kyphoplasty procedure (e.g., in the presence of active or incompletely treated local infection)
11. Positive baseline pregnancy test (for women of child-bearing potential)
12. Subject has neurologic deficit associated with the level(s) to be treated more severe than radiculopathy (e.g. myelopathy, cauda equina syndrome)
13. Subject has segmental kyphosis > 30° in area of treatment
14. Subject has uncontrolled coagulopathy
15. Subject cannot temporarily discontinue anticoagulation therapy
16. Subject has a known allergy to device materials / PMMA
17. Index VCF was exposed to high energy trauma
18. Subject has severe cardiopulmonary deficiencies as contra-indication to local or general anesthesia required for the procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05

PRIMARY OUTCOMES:
Improvement in functional status, as measured by the Oswestry Disability Index (ODI) | 1 month

SECONDARY OUTCOMES:
Change in Quality of Life (SF-35 Health Survey) | 1 month, 3 month
Change in Back Pain (VAS) | 1 month, 3 month
  Visual Analog Scale for pain
Change in Physical Disability associated with back pain (Roland-Morris Disability Questionnaire) | 1 month, 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vrionis, MD, MPH, PhD, Principal Investigator — H. Lee Moffitt Cancer Center